CLINICAL TRIAL: NCT00741221
Title: Pemetrexed Plus Bevacizumab in Pretreated, Advanced or Metastatic Non Small Cell Lung Cancer (NSCLC)
Brief Title: Pemetrexed Plus Bevacizumab in Non Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hellenic Oncology Research Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT/08.10
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Non-small-cell Lung Cancer
Keywords: Cancer; NSCLC; Docetaxel; Bevacizumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — Pemetrexed; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Pemetrexed/Bevacizumab
  Interventions: Drug: Pemetrexed; Drug: Bevacizumab

INTERVENTIONS:
Drug: Pemetrexed — Pemetrexed (IV) 500 mg/m2 on day 1 every 3 weeks for 6 cycles
  Other Names: Alimta
Drug: Bevacizumab — Bevacizumab (IV) 15 mgr/Kgr on day 1 every 3 weeks for 6 cycles After the end of the 6 cycles Bevacizumab will be administered alone at the dose of 15 mgr/Kgr (IV) every 3 weeks until disease progression
  Other Names: Avastin

SUMMARY:
This trial will evaluate the efficacy and safety of pemetrexed and bevacizumab combination in patients with pretreated, advanced non small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
Pemetrexed is and an effective and well tolerated cytotoxic agent in the 2nd line treatment of advanced or metastatic non small cell lung cancer (NSCLC). Recently, a phase III study of 1st line treatment in patients with advanced or metastatic NSCLC showed that the addition of bevacizumab to a platinum-based regimen provided a survival benefit. There are patients with NSCLC who have not received bevacizumab and have relapsed after 1st and/or 2nd line therapy. The evaluation of bevacizumab plus chemotherapy in such patients is justified. This study will evaluate the combination of pemetrexed and bevacizumab as 2nd or 3rd line treatment of NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed,
* Unresectable locally advanced (stage IIIB) or metastatic (stage IV) non-squamous NSCLC
* At least one and no more than two previous chemotherapy regimens for advanced - or metastatic NSCLC
* Measurable disease, defined as at least 1 bidimensionally measurable lesion ≥ 20 X 10 mm.
* Age ≥ 18 years.
* Performance status (WHO) 0-2.
* Life expectancy of at least 12 weeks.
* Adequate bone marrow (ANC ≥ 1,500/mm3, PLT ≥ 100,000/mm3, Hgb ≥ 11 g/dL), liver (Bilirubin ≤ 1.5 Upper normal limit, SGOT/SGPT ≤ 2.5 Upper normal limit in the absence of liver metastases or ≤ 5 Upper normal limit in the presence of liver metastases), and renal function (Creatinine ≤ 1,5 Upper normal limit).
* Patients must be able to understand the nature of this study and give written informed consent

Exclusion Criteria:

* Previous therapy with pemetrexed
* Second primary malignancy, except for non-melanoma skin cancer and in situ cervical cancer
* Pregnant or lactating women
* Any serious, uncontrolled comorbidity on the investigator's judgment. Uncontrolled infection
* Any sustained chronic toxicity > grade 2 according to the NCI CTCAE (version 3.0)
* Symptomatic neuropathy > grade 2 according to the NCI CTCAE (version 3.0)
* Brain metastases, except if radiated and asymptomatic
* Radiotherapy within the previous 4 weeks
* Previous radiotherapy to the only measurable lesion
* Proteinuria ≥ 500 mgr of protein daily
* Hemoptysis > 10 cc per event
* Clinically significant hematemesis
* Centrally located lesion or in contact with major vessels
* Pulmonary lesion with cavitation
* Documented hemorrhagic diathesis or coagulation disorder
* Cardiovascular disease (class II-IV NYHA congestive heart failure, myocardial infarction within the previous 4 months, unstable angina, LVEF < normal, ventricular arrhythmia, uncontrolled hypertension)
* Thrombotic event within the previous 6 months
* Concurrent use of aspirin > 325 mgr daily, low molecular weight heparin in therapeutic dose, warfarin or acenocoumarol, non-steroid anti-inflammatory agents
* Concurrent treatment with other anti-cancer drug
* Major surgical procedure within the previous 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-06; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 1 year

SECONDARY OUTCOMES:
Overall response rate | Objective responses confirmed by CT or MRI (on 3rd and 6th cycle)
Overall Survival | 1 year
Quality of life assessment | Assessment every two cycles
Toxicity profile | Assessment every two cycles

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Agelaki, MD, Principal Investigator — University Hospital of Crete, Dep of Medical Oncology; Manolis Kontopodis, MD, Principal Investigator — University Hospital of Crete
Locations (10):
- Greece (10):
  - University Hospital of Heraklion, Heraklion, Crete
  - University General Hospital of Alexandroupolis, Dep of Medical Oncology, Alexandroupoli
  - "Laikon" General Hospital, Medical Oncology Unit, Propedeutic Dep of Internal Medicine, Athens
  - 401 Military Hospital, Medical Oncology Unit, Athens
  - Air Forces Military Hospital, Dep of Medical Oncology, Athens
  - IASO" General Hospital of Athens, 1st Dep of Medical Oncology, Athens
  - Sismanogleio General Hospital, 1st, 2nd Dep of Pulmonary Diseases, Athens
  - Sotiria" General Hospital, 1st, 3rd, 8th Dep of Pulmonary Diseases, Athens
  - "Metaxa's" Anticancer Hospital of Piraeus,1st Dep of Medical Oncology, Piraeus
  - Theagenion" Anticancer Hospital of Thessaloniki, Thessaloniki